CLINICAL TRIAL: NCT03270098
Title: Improving Cognition Via Exercise in Schizophrenia
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Icahn School of Medicine at Mount Sinai (Other)
Collaborators: University of North Carolina, Chapel Hill (Other); Stanford University (Other); Augusta University (Other); Columbia University (Other); National Institute of Mental Health (NIMH) (NIH)
Responsible Party: Principal Investigator, David Kimhy, Associate Professor, Psychiatry, Icahn School of Medicine at Mount Sinai
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: GCO 17-1511; 1R01MH110623-01A1 (NIH); 3R01MH110623-03S1 (NIH)
Record Dates: First submitted 2017-08-30; First posted 2017-09-01 (Actual); Last update posted 2023-04-14 (Actual); Status verified 2023-04

CONDITIONS: Schizophrenia and Related Disorders
Keywords: Schizophrenia; Aerobic Exercise; Cognition; Daily Functioning; Biomarkers; Brain Derived Neurotrophic Factor; Suicide Risk
MeSH Terms: conditions — Schizophrenia | interventions — Exercise

STUDY DESIGN:
Intervention Model Description: This study is a single-blind, parallel assignment, multi-site randomized clinical trial designed to examine the impact of exercise on cognition, daily functioning, and biomarkers of cognitive change in people with schizophrenia.
Who Masked: Outcomes Assessor
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Aerobic Exercise (Experimental): Using trainer-led video calls with traditional callisthenic body movements (e.g., jumping jacks, burpees, etc.)
  Interventions: Behavioral: Aerobic Exercise
- Stretching and Toning Exercise (Active Comparator): Using trainer-led video calls with stretching and toning exercises.
  Interventions: Behavioral: Stretching and Toning Exercise

INTERVENTIONS:
Behavioral: Aerobic Exercise — Trainer-led one hour aerobic exercise sessions, three times per week, over 12 weeks.
  Arms: Aerobic Exercise
Behavioral: Stretching and Toning Exercise — Trainer-led one hour stretching-and-toning exercise sessions, three times per week, over 12 weeks.
  Arms: Stretching and Toning Exercise

SUMMARY:
People with schizophrenia display a broad range of cognitive impairments that have been identified as major determinants of poor functioning and disability. Also, people with schizophrenia are at increased risk for suicide, with approximately 40-50% of individuals attempting to take their own lives during their lifetime. The goal of the proposed study is to examine the impact of remote exercise training on cognition, suicide risk, daily functioning, and biomarkers of cognitive change and suicidality in people with schizophrenia.

DETAILED DESCRIPTION:
The goal of the proposed study is to examine the impact of remote exercise training on cognitive functioning in people with schizophrenia. People with schizophrenia display a broad range of cognitive impairments that have been identified as major determinants of poor functional outcome and disability, thus representing an important public health concern and a target for interventions. At present, available treatments offer only minimal to limited benefits to ameliorate these deficits. Extensive animal and human research literatures converge in supporting the positive influence of aerobic exercise training on cognitive functioning. Preliminary data indicate that aerobic exercise training is effective in improving cognitive functioning in people with schizophrenia. However, previous studies employed small samples, focused on a single or limited range of cognitive domains, and/or collected insufficient information on daily functioning or putative biomarkers underlying cognitive change. Supported by supplement funding from NIMH, the goal of the proposed study is also to explore the impact of remote exercise training on suicide risk in individuals with schizophrenia. People with schizophrenia are at increased risk for suicide, with approximately 40-50% of individuals attempting to take their own lives during their lifetime, and an estimated 5-10% actually being successful in completing suicide. This highly elevated risk represents a serious public health concern and an important target for interventions. However, available treatments offer only minimal to limited benefits to ameliorate this risk. Extensive animal and human research literatures converge in supporting the positive influence of AE training on a number of predictors of suicide risk including depressed mood, sleep difficulties, and poor cognition. Yet, at present there are no studies directly examining the impact of AE on suicide risk in this population.

ELIGIBILITY:
Inclusion Criteria:

* A DSM-V diagnosis of schizophrenia, schizoaffective, or schizophreniform disorder.
* Age 18-55 years.
* Taking antipsychotic medication for at least 8 weeks and on current doses for 4 weeks, and/or injectable depot antipsychotics with no change in the last 3 months.
* Capacity to understand all the potential risks and benefits of the study.
* Medically cleared by a physician to take part in VO2max tests and aerobic exercise training or stretching-and-toning exercise training.

Exclusion Criteria:

* A DSM-V diagnosis of alcohol/substance abuse (except nicotine) within the last month or a diagnosis of alcohol/substance dependence (except nicotine) within the last 6 months
* Initiation of anti-depressants, mood stabilizers, or other medications known to impact cognition in previous 4 weeks or any change in doses during this period.
* History of seizures/head trauma with loss of consciousness (>10 minutes) resulting in cognitive sequelae.
* Significant clinical abnormalities in physical examination, lab assessments, or ECG.
* Neurological/medical conditions that could interfere with study participation (e.g., unstable cardiac disease, stuttering).
* Body Mass Index (BMI) ≥ 40.
* Untreated hyper- or hypothyroidism.
* Being pregnant or nursing.
* Serious homicidal/suicidal risk (past 6 months).
* "Moderate" or more severe conceptual disorganization (PANSS≥4).
* Poor English reading ability (WTAR<7).
* Participation in a study with cognitive assessment in the past 3 months.
* Serious homicidal risk (past 6 months)

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 104 (Actual)
Dates: Start 2018-04-26 (Actual); Primary Completion 2023-01-31 (Actual); Study Completion 2023-01-31 (Actual)

PRIMARY OUTCOMES:
Change in the MATRICS Consensus Cognitive Battery (MCCB) | Baseline and 12 weeks
  The MCCB is a standardized battery designed to measure cognitive functioning in people with schizophrenia. The MCCB is represented as a composite T score. Change in the MCCB at 12 weeks as compared to baseline.
Change in VO2Max | Baseline and 12 weeks
  VO2Max (maximal oxygen consumption) is an index of the ability to consume oxygen and is a key indicator of aerobic fitness. Change in the VO2Max at 12 weeks as compared to baseline.

SECONDARY OUTCOMES:
Change in the Specific Levels of Functioning Scale (SLOF) | Baseline and 12 weeks
  The SLOF is a 43-item survey assessing multiple domains of daily functioning. Total score range from 43 to 215, with higher scores indicating better the overall functioning. Change in the SLOF at 12 weeks as compared to baseline.
Change in the UCSD Performance-based Skills Assessment (UPSA) | Baseline and 12 weeks
  The UPSA is performance-based measure of real-world daily functioning abilities. Participants receive scores for multiple domains, which are summed to create a summary score ranging from 0 to 100 with higher score indicating better overall functioning. Change in the UPSA at 12 weeks as compared to baseline.
Change in the Schizophrenia Cognition Rating Scale (SCoRS) | Baseline and 12 weeks
  The SCoRS is a 20-item clinician-administered interview assessing cognition-related daily functioning. Each item rated on a 4-point scale ranging from "no impairment" to "severe impairment". Total scores range from 20-80, with higher score indicating poorer functioning. Change in the SCoRS at 12 weeks as compared to baseline.
Serum BDNF | Baseline and 12 weeks
  BDNF is extracted from blood samples and serves as a biomarker of exercise-related cognitive changes. Change in the BDNF at 12 weeks as compared to baseline.
Change in Columbia Suicide Severity Rating Scale (C-SSRS) | Baseline and 12 weeks
  The C-SSRS is a semi-structured interview that measures 4 suicide risk related domains: ideation severity, ideation intensity, behavior, and lethality. Full scale from 1-10, with higher score indicating more suicidal ideation and behavior. Change in the C-SSRS at 12 weeks as compared to baseline.

CONTACTS AND LOCATIONS:
Overall Officials: David Kimhy, PhD, Principal Investigator — Icahn School of Medicine at Mount Sinai; T. Scott Stroup, MD, MPH, Principal Investigator — Columbia University
Locations (4):
- United States (4):
  - Stanford University, Stanford, California
  - Augusta University, Augusta, Georgia
  - Icahn School of Medicine at Mount Sinai, New York, New York
  - University of North Carolina, Chapel Hill, North Carolina

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Background] Kimhy D, Vakhrusheva J, Bartels MN, Armstrong HF, Ballon JS, Khan S, Chang RW, Hansen MC, Ayanruoh L, Lister A, Castren E, Smith EE, Sloan RP. The Impact of Aerobic Exercise on Brain-Derived Neurotrophic Factor and Neurocognition in Individuals With Schizophrenia: A Single-Blind, Randomized Clinical Trial. Schizophr Bull. 2015 Jul;41(4):859-68. doi: 10.1093/schbul/sbv022. Epub 2015 Mar 23. PMID 25805886
- [Background] Kimhy D, Lauriola V, Bartels MN, Armstrong HF, Vakhrusheva J, Ballon JS, Sloan RP. Aerobic exercise for cognitive deficits in schizophrenia - The impact of frequency, duration, and fidelity with target training intensity. Schizophr Res. 2016 Apr;172(1-3):213-5. doi: 10.1016/j.schres.2016.01.055. Epub 2016 Feb 3. No abstract available. PMID 26852401
- [Background] Kimhy D, Khan S, Ayanrouh L, Chang RW, Hansen MC, Lister A, Ballon JS, Vakhrusheva J, Armstrong HF, Bartels MN, Sloan RP. Use of Active-Play Video Games to Enhance Aerobic Fitness in Schizophrenia: Feasibility, Safety, and Adherence. Psychiatr Serv. 2016 Feb;67(2):240-3. doi: 10.1176/appi.ps.201400523. Epub 2015 Oct 1. PMID 26423100
- [Background] Armstrong HF, Bartels MN, Paslavski O, Cain D, Shoval HA, Ballon JS, Khan S, Sloan RP, Kimhy D. The impact of aerobic exercise training on cardiopulmonary functioning in individuals with schizophrenia. Schizophr Res. 2016 May;173(1-2):116-7. doi: 10.1016/j.schres.2016.03.009. Epub 2016 Mar 11. No abstract available. PMID 26976498
- [Background] Vakhrusheva J, Marino B, Stroup TS, Kimhy D. Aerobic Exercise in People with Schizophrenia: Neural and Neurocognitive Benefits. Curr Behav Neurosci Rep. 2016 Jun;3(2):165-175. doi: 10.1007/s40473-016-0077-2. Epub 2016 Apr 4. PMID 27766192
- [Background] Kimhy D, Vakhrusheva J, Bartels MN, Armstrong HF, Ballon JS, Khan S, Chang RW, Hansen MC, Ayanruoh L, Smith EE, Sloan RP. Aerobic fitness and body mass index in individuals with schizophrenia: Implications for neurocognition and daily functioning. Psychiatry Res. 2014 Dec 30;220(3):784-91. doi: 10.1016/j.psychres.2014.08.052. Epub 2014 Sep 3. PMID 25219618
- [Background] Ospina LH, Wall M, Jarskog LF, Ballon JS, McEvoy J, Bartels MN, Buchsbaum R, Sloan RP, Stroup TS, Kimhy D. Improving Cognition via Exercise (ICE): Study Protocol for a Multi-Site, Parallel-Group, Single-Blind, Randomized Clinical Trial Examining the Efficacy of Aerobic Exercise to Improve Neurocognition, Daily Functioning, and Biomarkers of Cognitive Change in Individuals with Schizophrenia. J Psychiatr Brain Sci. 2019;4:e190020. doi: 10.20900/jpbs.20190020. Epub 2019 Dec 30. PMID 31938726
- [Derived] Beck-Felts K, Goodman M, Ospina LH, Wall M, McEvoy J, Jarskog LF, Ballon JS, Bartels MN, Buchsbaum R, Sloan RP, Stroup TS, Kimhy D. Suicide Reduction in Schizophrenia via Exercise (SUnRISE): study protocol for a multi-site, single-blind, randomized clinical trial of aerobic exercise for suicide risk reduction in individuals with schizophrenia. Trials. 2020 Oct 21;21(1):871. doi: 10.1186/s13063-020-04788-z. PMID 33087170